CLINICAL TRIAL: NCT03641755
Title: A Phase Ib/II Study of Olaparib With Sapacitabine in BRCA Mutant Breast Cancer
Brief Title: Olaparib + Sapacitabine in BRCA Mutant Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: AstraZeneca (Industry); Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Filipa Lynce, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-223
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sapacitabine; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level -1: Sapacitabine (100 mg) + Olaparib (300 mg) (Experimental): * Olaparib will be administered orally twice daily for each 28-day cycle
  * Sapacitabine will be administered orally once daily on days 1 - 5 and 8 - 12 of every 28-day cycle
  Interventions: Drug: Sapacitabine; Drug: Olaparib
- Dose Level 1: Sapacitabine (150 mg) + Olaparib (300 mg) (Experimental): * Olaparib will be administered orally twice daily for each 28-day cycle
  * Sapacitabine will be administered orally once daily on days 1 - 5 and 8 - 12 of every 28-day cycle
  Interventions: Drug: Sapacitabine; Drug: Olaparib
- Dose Level 2: Sapacitabine (200 mg) + Olaparib (300 mg) (Experimental): * Olaparib will be administered orally twice daily for each 28-day cycle
  * Sapacitabine will be administered orally once daily on days 1 - 5 and 8 - 12 of every 28-day cycle
  Interventions: Drug: Sapacitabine; Drug: Olaparib
- Dose Level 3: Sapacitabine (250 mg) + Olaparib (300 mg) (Experimental): * Olaparib will be administered orally twice daily for each 28-day cycle
  * Sapacitabine will be administered orally once daily on days 1 - 5 and 8 - 12 of every 28-day cycle
  Interventions: Drug: Sapacitabine; Drug: Olaparib

INTERVENTIONS:
Drug: Sapacitabine — Sapacitabine may help to stop the growth of some types of cancers
  Other Names: CYC682
Drug: Olaparib — Olaparib is an inhibitor of PARP (poly [adenosine diphosphate-ribose] polymerase), which means that it stops PARP from working
  Other Names: Lynparza

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for breast cancer with a BRCA mutation.

The interventions involved in this study are:

* Sapacitabine (CYC682)
* Olaparib (Lynparza™)

DETAILED DESCRIPTION:
This is a Phase I/II clinical trial. A Phase I clinical trial tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied. It also means that the FDA (the U.S. Food and Drug Administration) has not approved the combination of Olaparib and Sapacitabine as a treatment for any disease.

The FDA (the U.S. Food and Drug Administration) has approved Olaparib as a treatment for metastatic HER2 negative breast cancer with a BRCA mutation. Olaparib is an inhibitor of PARP (poly [adenosine diphosphate-ribose] polymerase), which means that it stops PARP from working. PARP is an enzyme (a type of protein) found in the cells of the body. In normal cells when DNA is damaged, PARP helps to repair the damage.

The FDA has not approved Sapacitabine for use in patients including people with this type of cancer. Sapacitabine and drugs of its class have been shown to have antitumor properties in many types of cancer, e.g., leukemia, lung, breast, ovarian, pancreatic and bladder cancer. Sapacitabine may help to stop the growth of some types of cancers.

In this research study, the investigators are evaluating the safety and effectiveness of Olaparib in combination with Sapacitabine in BRCA mutant breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer that is metastatic or unresectable.
* Documented germline mutation in BRCA1 or BRCA2 that is predicted to be deleterious or suspected deleterious (known or predicted to be detrimental/lead to loss of function). Testing may be completed by any CLIA-certified laboratory.
* Patients with estrogen and/or progesterone receptor-positive disease must have received and progressed on at least one endocrine therapy (adjuvant or metastatic), or have disease that the treating physician believes to be inappropriate for endocrine therapy.
* Patients with HER2-positive disease must have received and progressed on two lines of HER2-directed therapy in the metastatic setting.
* Age ≥ 18 years
* ECOG performance status of 0-1 (please see Appendix A).
* Participants enrolling to the phase I portion of the study must have evaluable or measurable disease; participants enrolling to the phase II portion of the study must have measurable disease per RECIST 1.1 criteria (please see Section 11).
* Adequate organ and bone marrow function as defined below:

  * Hemoglobin ≥ 10 g/dL
  * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L
  * Platelet count ≥ 100 × 109/L
  * Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
  * AST(SGOT) / ALT (SGPT) ≤ 2.5 × institutional ULN, OR
  * AST(SGOT) / ALT (SGPT) ≤ 5 × institutional ULN if liver metastases are present
  * Creatinine Clearance estimated (using the Cockcroft-Gault equation) of ≥ 51 mL/min
* Ability to understand and willingness to sign an informed consent document.
* Ability to swallow and retain oral study medication.
* Female participants must be postmenopausal or must have a negative serum pregnancy test performed during screening. Postmenopausal is defined as:

  * Amenorrhoeic for 1 year or more following cessation of exogenous hormonal treatments
  * Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the postmenopausal range for women under 50.
  * Radiation-induced oophorectomy with last menses >1 year ago
  * Chemotherapy-induced menopause with >1 year interval since last menses
  * Status post surgical sterilization (bilateral oophorectomy or hysterectomy)
* The effects of sapacitabine and olaparib on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use two highly effective forms of contraception for the duration of study participation and 6 months after the last dose of sapacitabine and/or olaparib. Men must agree to use two highly effective forms of contraception for the duration of study participation and 3 months after the last dose of sapacitabine and/or olaparib. A list of acceptable methods is listed in Section 5.5.3.4.
* Participants must be willing and able to comply with the protocol for the duration of the study, including undergoing treatment and scheduled visits and examinations.
* Participants enrolling to the phase II portion of the trial must be willing to undergo a biopsy at baseline; if their disease is not accessible for biopsy they are still eligible to participate.

Exclusion Criteria:

* Any previous treatment with a PARP inhibitor, including but not limited to olaparib.
* Any previous treatment with sapacitabine.
* Patients who have had prior systemic chemotherapy, immune therapy, or investigational therapy within 3 weeks of study entry. Endocrine therapy must have been discontinued at least 7 days prior to Cycle 1 Day 1. Patients may receive bisphosphonates or denosumab during the study.
* Patients who have received prior radiotherapy within 1 week of study entry.
* Participants with active pneumonitis.
* Patients who have undergone major surgery or have ongoing persistent toxicities within 2 weeks prior to study entry. Patients must have recovered to baseline or ≤ Grade 1 from any effects of any major surgery prior to study entry with the exception of any grade of alopecia and persistent grade ≤ 2 peripheral neuropathy
* For enrollment during phase II: patients who have received more than 3 prior lines of cytotoxic chemotherapy for metastatic disease. Prior treatments with hormonal therapy and non-hormonal targeted therapy are allowed and not counted as a prior line of cytotoxic chemotherapy. For the purposes of this protocol, the combination of an aromatase inhibitor and everolimus is not considered cytotoxic chemotherapy.
* Patients with a history of treated central nervous system (CNS) metastases are eligible, provided they meet all of the following criteria:

  * Disease outside the CNS is present
  * No clinical evidence of progression in the CNS since completion of CNS-directed therapy
  * Minimum of 2 weeks between completion of radiotherapy and Cycle 1 Day 1
  * Recovery from significant (≥ Grade 3) acute toxicity with no requirement for escalating doses of corticosteroid over the 7 days prior to treatment start.
  * Participants requiring concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to study entry is 2 weeks.
* Participants requiring concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to study entry is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Participants with a QTcF of >470 msec on screening ECG.
* Participants with a personal or family history of long QT syndrome.
* Pregnant women are excluded from this study because olaparib and sapacitabine are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study agents, breastfeeding should be discontinued if the mother is treated with olaparib or sapacitabine and for one month after receiving the last dose.
* Participants with known active Hepatitis B, C, or known HIV positive status.
* Participants unable to swallow orally administered medication and participants with gastrointestinal disorders that are likely to interfere with absorption of the study medications in the opinion of the treating investigator (e.g. malabsorption syndrome or major stomach or bowel resections).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sapacitabine or olaparib.
* Patients with a history of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
* History of a previous allogeneic bone marrow transplant or double umbilical cord blood transplantation.
* Patients with a history of a second primary malignancy, with the following exceptions: adequately treated non-melanoma skin cancers, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS) of the breast, stage 1 grade 1 endometrial carcinoma, and any other solid tumor or lymphoma (without bone marrow involvement) diagnosed ≥ 5 years prior to study entry and treated with no evidence of disease recurrence; other exceptions may exist following agreement with the principal investigator who believes disease recurrence is unlikely.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants who are involved in the planning and/or conduct of the study (applies to both pharmaceutical company staff and/or staff at the study site).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2026-10-22 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Assessed from the time of the first patient registration to the time that the last patient comes off protocol therapy in the dose escalation phase, up to 41 months
  The dose level immediately below the maximally-administered dose (MAD; defined as the dose level where at least two participants develop dose-limiting toxicity [DLT]) will be defined as the MTD. In the situation where none of the dose levels have ≥ 2 DLTs, the MTD will be the highest dose administered. The MTD will be established in a minimum of 6 participants.
Recommended Phase II dose (RPIID) | Assessed from the time of the first patient registration to the time that the last patient comes off protocol therapy, up to 41 months
  The highest dose level below the MAD at which ≤1 out of 6 patients develop DLT. The RPIID will be established in a minimum of 6 participants.
Objective Response Rate | Assessed for each patient from the time of registration until 30 days after removal from protocol therapy or until death, whichever occurs first, up to 41 months
  Defined as the percentage of patients achieving a complete response (disappearance of all target and non-target lesions; no new lesions) or partial response (at least 30% decrease in the sum of the diameters of target lesions; persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits ["non-CR/non-PD" in non-target lesions]; and no new lesions) based on RECIST 1.1

SECONDARY OUTCOMES:
Progression-Free Survival | Assessed for each patient from the time of registration until 30 days after removal from protocol therapy or until death, whichever occurs first, up to 41 months
  Defined as the time from registration to the earlier of progression by RECIST 1.1 or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation.
Dose Limiting Toxicity | Assessed for each patient from the start of protocol therapy to the end of the first cycle of therapy (28 days post start of therapy)
  Evaluated among participants enrolled to the phase I trial during the first cycle of therapy. DLTs are defined as toxicities that are considered at least possibly related to the study regimen and that fit one or more of the following criteria:
  * Any death not clearly due to the underlying disease or extraneous causes
  * Any non-hematologic toxicity ≥ Grade 3
  * Any occurrence of Hy's Law (see protocol Appendix B)
  * Febrile neutropenia ≥ Grade 3
  * Grade 4 neutropenia or thrombocytopenia lasting >7 days
  * Thrombocytopenia with bleeding ≥ Grade 3
  * ≥ Grade 3 nausea, vomiting, diarrhea lasting > 72 hours with adequate antiemetic or other supportive care.
  * ≥ Grade 3 fatigue lasting > 7 days
  * ≥Grade 3 electrolyte abnormality that lasts > 72 hours with no clinical symptoms.
  * ≥ Grade 3 electrolyte abnormality with clinical symptoms, regardless of duration.
  Toxicities are defined according to NCI CTCAE, Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Filipa Lynce, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Broad Institute of MIT, Cambridge, Massachusetts

IPD SHARING:
Plan to Share IPD: No